CLINICAL TRIAL: NCT05983926
Title: To Explore the Efficacy and Safety of Surgical Treatment for Constipation, as Well as the Changes of Postoperative Intestinal Motility, Flora, Nutritional Status and Other Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, Clinical Professor, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STC-20230704
Record Dates: First submitted 2023-07-03; First posted 2023-08-09 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Constipation; Surgical Treatment
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Differences in conditions before and after surgical treatment of constipation (Experimental)
  Interventions: Procedure: Subtotal colectomy was performed

INTERVENTIONS:
Procedure: Subtotal colectomy was performed — Colonic subtotal resection, also known as subtotal colectomy, is a surgical procedure used to treat colonic diseases such asconstipation, colon cancer, ulcerative colitis, and others.
  The purpose of this surgery is to remove a portion of the colon in the patient's body. Unlike a total colectomy, which involves removing the entire colon, a subtotal colectomy only removes a portion of the colon. The procedure typically involves removing the diseased part of the colon and reconnecting the remaining colon. This allows for the preservation of some normal colonic function, enabling the patient to have regular bowel movements.

SUMMARY:
Chronic constipation is a heterogeneous disease with multiple symptoms, and its incidence is on the rise in many countries. It has become a common disease affecting the quality of life. When these patients fail to respond to standardized and systematic non-surgical treatment, and the relevant examination suggests that there are surgical indications, surgical treatment should be considered. TThe objective of this study was to explore the efficacy and safety of surgical treatment for constipation, as well as the changes in postoperative nutrition, intestinal motility, intestinal flora and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Disease duration more than 6 years;
* Wexner constipation score >15;
* No response to medical treatment, biofeedback and fecal microbiota transplantation;
* according to the surgical indications;
* All patients were informed of this study and signed the informed consent.

Exclusion Criteria:

* Suffering from mental disorders or cognitive impairment;
* With malignant tumors; -
* With history of gastrointestinal surgery;
* Complicated with other organ dysfunction;
* With immune system diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The nutritional status of the patients was assessed according to the scores of nutritional risk screening and assessment tool Nutritional Risk Screening2022（NRS2002) | Baseline and 1、6、12 and 24 months after surgery
  The full length of NRS2002 is called Nutritional Risk Screening2022. The minimum score is 0 and the maximum score is 3, with higher scores indicating higher nutritional risk.
The nutritional status of the patients was assessed according to the scores of nutritional risk screening and assessment tool Malnutrition Universal Screening Tool （MUST). | Baseline and 1、6、12 and 24 months after surgery
  The full name of MUST is Malnutrition Universal Screening Tool, score 0: low risk; Score 1: moderate risk; A score of 2 or higher is considered high risk.
The nutritional status of the patients was assessed according to the scores of nutritional risk screening and assessment tool Mini Nutritional Assessment （MNA). | Baseline and 1、6、12 and 24 months after surgery
  Mini Nutritional Assessment (MNA) is defined as "good nutritional status" when MNA≥24. 17≤MNA < 24, nutritional risk; MNA < 17 indicated malnutrition.
The peristalsis status of patients was evaluated according to the frequency of defecation and the character of feces. | Baseline and 1、6、12 and 24 months after surgery
The changes of fecal microbiota were detected by 16SDNA sequencing. | Baseline and 1、6、12 and 24 months after surgery
Quantitative changes in immune cells were determined by flow cytometry of blood samples. | Baseline and 1、6、12 and 24 months after surgery
Changes of intestinal motility after surgical treatment for constipation. | Baseline and 1、6、12 and 24 months after surgery
  The intestinal transit time of patients was detected
Changes of defecation after surgical treatment for constipation. | Baseline and 1、6、12 and 24 months after surgery
  The frequency of postoperative defecation, the characteristics of stool and the force of defecation were studied by asking patients to record their defecation diary.
Changes of quality of life after surgical treatment for constipation. | Baseline and 1、6、12 and 24 months after surgery
  Patients were evaluated using the quality of Life assessment scale.

CONTACTS AND LOCATIONS:
Overall Officials: Le Wang, Master, Principal Investigator — Intestinal Microenvironment Treatment Center of General Surgery, Shanghai Tenth People's Hospital, Tenth People's Hospital of Tongji University
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided